CLINICAL TRIAL: NCT02043639
Title: A Study of Effectiveness of clinicCompanion. Compared to the Use of a Goniometer for Range of Motion Measurement.
Brief Title: ClinicCompanion. Compared to the Use of a Goniometer
Status: Terminated | Type: Observational
Why Stopped: Change in technology
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Medical Companion LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 13-40 ClinicCompanion.
Record Dates: First submitted 2014-01-14; First posted 2014-01-23 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2016-04

CONDITIONS: Shoulder Impingement Syndrome
Keywords: rotation; shoulder; joint; ROM; abduction,; internal rotation,; external rotation,; flexion; normal; joint movement; physical examination
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this study, the goal is to find out if the clinicCompanion™ is effective in measuring range of motion when compared to the goniometer. Currently, the goniometer is an approved device to measure range of motion by the FDA, but the clinicCompanion™ is not.

DETAILED DESCRIPTION:
The study procedure will test the range of motion of the subjects shoulders two different ways: using a goniometer and using the clinicCompanion™. Both tools are designed to measure the degree of movement subjects are able to do. Researchers will take 12 measurements on each arm for each device, for a total of 24 measurements per device. That is a total of 48 measurements for both devices.

ELIGIBILITY:
Inclusion Criteria:

* new or established clinic patients from PI's medical practice at Aurora St. Luke's Medical Center
* 18 years of age and older

Exclusion Criteria:

* no use of limbs
* amputees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New or established clinic patients from Aurora St. Luke's Medical Center. The subjects will be recruited from the principal investigator's medical practice. Any patient may be included in the study, regardless of his/her diagnosis and must be 18 years of age and older.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Control cost and enhance accuracy of measurement | The goal is to recruit 75 subjects in 18 months
  By freeing the doctor from data collection, he or she will be able to spend more time with patient discussing medical conditions and providing pertinent information

CONTACTS AND LOCATIONS:
Overall Officials: Maharaj m Singh, PHD, Principal Investigator — Wake Forest University Health Sciences; Navjot m Kohli, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora St Lukes Medical Center, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Mullaney MJ, McHugh MP, Johnson CP, Tyler TF. Reliability of shoulder range of motion comparing a goniometer to a digital level. Physiother Theory Pract. 2010 Jul;26(5):327-33. doi: 10.3109/09593980903094230. PMID 20557263
- [Background] van de Pol RJ, van Trijffel E, Lucas C. Inter-rater reliability for measurement of passive physiological range of motion of upper extremity joints is better if instruments are used: a systematic review. J Physiother. 2010;56(1):7-17. doi: 10.1016/s1836-9553(10)70049-7. PMID 20500132
- [Background] MacDermid JC, Chesworth BM, Patterson S, Roth JH. Intratester and intertester reliability of goniometric measurement of passive lateral shoulder rotation. J Hand Ther. 1999 Jul-Sep;12(3):187-92. doi: 10.1016/s0894-1130(99)80045-3. PMID 10459526
- [Background] Riddle DL, Rothstein JM, Lamb RL. Goniometric reliability in a clinical setting. Shoulder measurements. Phys Ther. 1987 May;67(5):668-73. doi: 10.1093/ptj/67.5.668. PMID 3575423
- [Background] Khoshelham K, Elberink SO. Accuracy and resolution of Kinect depth data for indoor mapping applications. Sensors (Basel). 2012;12(2):1437-54. doi: 10.3390/s120201437. Epub 2012 Feb 1. PMID 22438718
- [Background] Dutta T. Evaluation of the Kinect sensor for 3-D kinematic measurement in the workplace. Appl Ergon. 2012 Jul;43(4):645-9. doi: 10.1016/j.apergo.2011.09.011. Epub 2011 Oct 20. PMID 22018839